CLINICAL TRIAL: NCT02050477
Title: Laparoscopic Non Banded Vertical (Magenstrasse and Mill) Gastroplasty In Bariatric Surgery. Morbidity and Results on Weight Loss and Associated Co-morbidities
Brief Title: Clinical Study of Laparoscopic Non Banded Vertical Gastroplasty in Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Arnaud De Roover, Professeur de Clinique, Chef de Clinique, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B707201214181
Record Dates: First submitted 2014-01-25; First posted 2014-01-30 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: Obesity; Bariatric; Surgery; Sleeve; Gastroplasty; Laparoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopic Vertical Gastroplasty (Experimental)
  Interventions: Procedure: Laparoscopic Vertical Gastroplasty

INTERVENTIONS:
Procedure: Laparoscopic Vertical Gastroplasty — The Magenstrasse and Mill procedure is a conservative vertical gastroplasty described in 1987 through a laparotomy. A tubular gastric pouch is created by a vertical stapling extending from the antrum to the angle of Hiss. In this study, we evaluate the laparoscopic technique of the procedure.

SUMMARY:
Evaluation of the laparoscopic approach of the Magenstrasse and Mill procedure in a prospective study of 100 patients

DETAILED DESCRIPTION:
The laparoscopy is performed under general anesthesia with a 5 ports access under 14mm Hg pressure. After opening of the gastrocolic ligament and division of any adhesions between stomach and pancreas a circular opening is performed at the junction of corpus and antrum of the stomach with a circular stapler. A tubular gastric pouch is then created along a calibration tube at the lesser curvature by a vertical stapling starting from the circular opening to the angle of Hiss.

ELIGIBILITY:
Inclusion Criteria:

* Assessment by a multidisciplinary team specialized in bariatric and metabolic surgery including surgeon, endocrinologist, psychologist and/or psychiatrist, dietician
* BMI>40
* BMI>35 with diabetes or sleep apnea syndrome or hypertension treated with 3 drugs for at least one year
* Male or female patients between 18 and 75 years of age; fertile female patients must use a reliable contraception method;
* No previous bariatric procedure
* Informed consent given by patient

Exclusion Criteria:

* Medical contra-indication for a general anesthesia, or abdominal surgery (allergies to anesthetic drugs, cardio-vascular, pulmonary, or renal conditions leading to an unacceptable risk for the procedure
* Psychological-Psychiatric (boulimia, severe depression, psychotic condition)
* Non stabilized endocrine disorder, with potential interference on weight and/or diabetic condition
* Unability to understand goal of the study, plan of treatment and follow-up
* Large hiatal hernia and/or severe esophageal reflux disease
* Grazer, Sweet eater behavior

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Morbidity/Mortality | 1 month
Effect of the procedure on weight loss | 1 year
  Evaluation at 1,3,6 and 12 months through clinical evaluation.

SECONDARY OUTCOMES:
Reflux disease | 1 year
  Evaluation at 1,3,6 and 12 months through clinical evaluation, Gastroscopy if symptoms present. Upper GI opacification at one year will be performed for all patients.
Effect of procedure on obesity associated co-morbidities | 1 year
  Co-morbidities include diabetes, hypertension, sleep apnea syndrome, dyslipemia Evaluation at 1,3,6 and 12 months through clinical evaluation and blood assessment

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud De Roover, MD, Principal Investigator — Dept of Abdominal Surgery and Transplantation CHU Liège Belgium
Locations (1):
- Dept of Abdominal Surgery and Transplantation, CHU Liège, Liège, Liège, Belgium